CLINICAL TRIAL: NCT00635167
Title: Contrast Enhanced Transrectal Ultrasound (TRUS) to Assess Prostatic Vascularity as a Measure of Treatment Response and Early Prediction of Treatment Failure After XRT
Brief Title: Contrast Enhanced Transrectal Ultrasonography (TRUS) to Assess Prostatic Vascularity After Radiotherapy (XRT)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by PI final report submitted
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07D.218; JT 1259 (Other: JeffTrial Number)
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; prostatic vascularity; External Beam Radiation treatment; Contrast Enhanced transrectal Ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contrast Enhanced Transrectal Ultrasound (TRUS) (Experimental)
  Interventions: Drug: Contrast Enhanced-Transrectal Ultrasound

INTERVENTIONS:
Drug: Contrast Enhanced-Transrectal Ultrasound — Drug Once a subject is identified TRUS schedule will be set up revolving around the EBRT treatment schedule. A schedule of 6 contrast enhanced TRUS examinations per subject is planned as follows: week 0 (prior to EBRT, baseline [Visit 2]); week 5 (middle of treatment [Visit 3]); week 10 (end of treatment [Visit 4]); week 18 (2 months after end of EBRT [Visit 5]); week 26 (4 months after end of EBRT [Visit 6]); and week 36 (6 months after end of EBRT [Visit 7]).

SUMMARY:
Solid tumors, including prostate cancer, commonly exhibit tumor-associated neovascularity (growth of new blood vessels to feed the tumor) with increased microvessel density. Systemic, hormonal, and radiotherapy treatments typically decrease or suppress tumor - associated vascularity through several mechanisms, including apoptosis (process of cell death) and anti-angiogenic pathways (ways to destroy new blood vessel growth). Previously at the investigators' center, they have demonstrated that increased prostatic vascularity (blood vessels defined to prostate) detected ultrasonographically correlated with disease free survival after radical prostatectomy (surgical removal of entire prostate), and may be indicative of higher grade, higher stage disease. The significance of prostate neovascularity in response to treatment with external beam radiotherapy (EBRT) (standard of care) has not been well studied. The investigators hypothesize that prostate cancer that recurs after radiotherapy may exhibit measurable patterns of tumor-associated vascularity, which may represent a minimally invasive marker of cancer stage, grade and response to treatment. The investigators propose a pilot study to assess the feasibility of serial enhanced transrectal ultrasonography (TRUS) examinations during and after radiotherapy for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40 - 80 years old
* Biopsy proven intermediate/high risk clinically localized prostate cancer, as determined by a Gleason score of 7 or higher, clinical stage T2b or higher, or PSA > 10. Pathology will be confirmed by at least two reviews
* Patients opting for EBRT (external beam radiation therapy, standard of care) without hormonal ablation
* Ability to undergo serial TRUS procedures
* Ability to give informed consent

Exclusion Criteria:

* Subject has known hypersensitivity to octafluoropropane.
* Evidence of distant metastatic disease on staging evaluation
* Previous treatment for prostate cancer, including any form of androgen ablation
* Previous procedures involving the anus or rectum, making serial TRUS difficult or dangerous
* Expected life expectancy less than 10 years
* Baseline testosterone < 200 ng/dL
* Subject with cardiac shunts and elevated pulmonary hypertension
* Subject has worsening or clinically unstable congestive heart failure.
* Subject has acute myocardial infarction or acute coronary syndrome.
* Subject has ventricular arrhythmias or is high risk for arrhythmias.
* Subject has respiratory failure, severe emphysema or pulmonary emboli.
* Subject has a history of cardiac shunt or pulmonary hypertension.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2011-05-12 (Actual); Study Completion 2011-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edouard J Trabulsi, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Halpern EJ, Frauscher F, Strup SE, Nazarian LN, O'Kane P, Gomella LG. Prostate: high-frequency Doppler US imaging for cancer detection. Radiology. 2002 Oct;225(1):71-7. doi: 10.1148/radiol.2251011938. PMID 12354987
- [Background] Halpern EJ, Frauscher F, Rosenberg M, Gomella LG. Directed biopsy during contrast-enhanced sonography of the prostate. AJR Am J Roentgenol. 2002 Apr;178(4):915-9. doi: 10.2214/ajr.178.4.1780915. PMID 11906872
- [Background] Nelson ED, Slotoroff CB, Gomella LG, Halpern EJ. Targeted biopsy of the prostate: the impact of color Doppler imaging and elastography on prostate cancer detection and Gleason score. Urology. 2007 Dec;70(6):1136-40. doi: 10.1016/j.urology.2007.07.067. PMID 18158034
- [Background] Linden RA, Halpern EJ. Advances in transrectal ultrasound imaging of the prostate. Semin Ultrasound CT MR. 2007 Aug;28(4):249-57. doi: 10.1053/j.sult.2007.05.002. PMID 17874649
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contrast Enhanced Transrectal Ultrasound (TRUS)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Contrast Enhanced Transrectal Ultrasound (TRUS)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Measurable Decrease in Prostate Vascularity During and/or After Radiation Treatment
Time Frame: 1 year
Population: This trial did not accrue well and was terminated prematurely. No data were not collected or analyzed.
Arm/Group | Contrast Enhanced Transrectal Ultrasound (TRUS)
Number analyzed (Participants) | 0

2. Secondary Outcome: Sonographic Appearance of Prostate and Prostate Vascularity Before, During and After External Beam Radiotherapy (Standard of Care) for Prostate Cancer
Time Frame: 1 year
Population: This trial did not accrue well and was terminated prematurely. No data were not collected or analyzed.
Arm/Group | Contrast Enhanced Transrectal Ultrasound (TRUS)
Number analyzed (Participants) | 0

3. Secondary Outcome: Patient Tolerance of TRUS Evaluation During/After Radiation Treatment
Time Frame: 1 year
Population: This trial did not accrue well and was terminated prematurely. No data were not collected or analyzed.
Arm/Group | Contrast Enhanced Transrectal Ultrasound (TRUS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Contrast Enhanced Transrectal Ultrasound (TRUS)
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes